CLINICAL TRIAL: NCT05362773
Title: A Phase 1, First-in-Human, Dose Escalation Study of MGD024, a CD123 x CD3 Bispecific DART Molecule, in Patients With Select Relapsed or Refractory Hematologic Malignancies
Brief Title: A Study of MGD024 in Patients With Relapsed or Refractory Hematologic Malignancies
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: MacroGenics (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: CP-MGD024-01
Record Dates: First submitted 2022-05-02; First posted 2022-05-05 (Actual); Last update posted 2026-01-13 (Actual); Status verified 2026-01

CONDITIONS: Leukemia, Acute Myeloid; Myelodysplastic Syndromes; Classical Hodgkin Lymphoma; Leukemia, B-cell; Leukemia, Hairy Cell; Mastocytosis, Aggressive Systemic; Blastic Plasmacytoid Dendritic Cell Neoplasm; Chronic Myeloid Leukemia
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Myelodysplastic Syndromes; Leukemia, B-Cell; Leukemia, Hairy Cell; Mastocytosis, Systemic; Blastic Plasmacytoid Dendritic Cell Neoplasm; Leukemia, Myelogenous, Chronic, BCR-ABL Positive

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Dose Escalation (Experimental): Escalating doses of MGD024 will be assigned based on safety and tolerability of the previous dose level.
  Interventions: Drug: MGD024

INTERVENTIONS:
Drug: MGD024 — MGD024 is a CD123 x CD3 bispecific DART® molecule designed to target CD123-expressing leukemic cells for elimination by CD3-expressing T lymphocytes.

SUMMARY:
CP-MGD024-01 is a Phase 1, open-label, multi-center study of MGD024 as a single agent in participants with select blood cancers that have not responded to treatment with standard therapies or who have relapsed after treatment. The study is designed to determine the safety, tolerability, pharmacokinetics (affect of the body on the drug), pharmacodynamic (affect of the drug on the body), immunogenicity (development of antibodies against the drug), and preliminary anti-cancer effect of MGD024.

Participants will receive treatment with MGD024 in consecutive 28-day cycles for a study treatment period of up to 12 cycles (approximately 1 year) or until treatment or study discontinuation criteria are met. Response assessments will be performed after Cycle 1 and then after every even numbered cycle starting with Cycle 2 until progression or study treatment discontinuation. Participants will be checked for side effects throughout the study.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients at least 18 years of age, able to provide informed consent and willing to comply with all study procedures.
* Participants with

  * primary or secondary acute myeloid leukemia (AML) except acute promyelocytic leukemia,
  * primary or secondary myelodysplastic syndrome (MDS) with prognostic score of >3 and <20% bone marrow blasts,
  * classical Hodgkin lymphoma (cHL),
  * chronic myelogenous leukemia (CML),
  * b-cell acute lymphocytic leukemia (B-ALL),
  * hariy cell leukemia (HCL),
  * advanced systemic mastocytosis (ASM), or
  * blastic plasmacytoid dendritic cell neoplasm (BPDCM)
* Relapsed after or refractory to at least one prior line of therapy and with no available potentially curative treatment option.
* Evidence of at least 20% of malignant cells with CD123 expression.
* Eastern Cooperative Oncology Group (ECOG) performance status of ≤ 2.
* Life expectancy of at least 12 weeks.
* Acceptable laboratory values, and heart function.
* Continuing side effects of prior treatment are mild
* Women and men of childbearing potential must agree to use highly effective forms of contraception throughout the study through 4 months after the last dose of MGD024.

Exclusion Criteria:

* Prior treatment with an anti-CD123-directed agent (except patients with BPDCN, who are allowed to have received prior tagraxofusp).
* Known involvement of central nervous system (CNS) by the disease under investigation.
* History or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the trial, interfere with the patient's participation for the full duration of the trial, or is not in the best interest of the patient.
* Systemic anti-cancer therapy, investigational therapy, corticosteroids or other immune suppressive drugs within 14 days of first dose
* Vaccination with any live virus vaccine within 4 weeks prior to first dose. Inactivated annual influenza and SARS-CoV-2 vaccination are allowed.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 130 (Estimated)
Dates: Start 2022-07-13 (Actual); Primary Completion 2026-11 (Estimated); Study Completion 2027-05 (Estimated)

PRIMARY OUTCOMES:
Number of severe side effects in patients receiving MGD024 | First 28 days of the study
  Observation of side effects determines the highest safe dose for further study
Number and types of adverse events (AEs), including serious adverse events (SAEs), and AEs leading to treatment discontinuation. | Throughout study participation, up to 12 months.
  Observation of side effects determines the highest safe dose for further study

SECONDARY OUTCOMES:
Mean maximum concentration | Throughout study participation, up to 12 months.
  The highest concentration of MGD024 at the end of the infusion
Mean area under the concentration-time curve (AUC) | Throughout study participation, up to 12 months.
  Total body exposure to MGD024
Number of participants with anti-drug antibody formation | Throughout study participation, up to 12 months.
  Number of patients who develop antibodies against MDG024
Overall response rate | Disease response assessment on Day 28, Day 56, then every 56 days throughout the study, up to 12 months.
  The proportion of patients with a complete response or a partial response to treatment
Complete response rate | Disease response assessment on Day 28, Day 56, then every 56 days throughout the study, up to 12 months.
  The proportion of patient achieving a complete response according to disease-specific criteria
Median progression free survival | Disease response is assessed approximately every 56 days throughout the study, up to 12 months.Assessed from Day 1 throughout the study until individual participant discontinuation, up to 12 months. Survival from Day 1 throughout the study.
  The time between the first dose date to the date of first documented disease-specific progression or death from any cause
Median time to response | Disease response is assessed approximately every 56 days throughout the study, up to 12 months.
  The time between the first dose and the date of complete or partial response.
Median duration of response | Disease response is assessed approximately every 56 days throughout the study, up to 12 months.
  The time between the date of initial response to the date of disease-specific progression or death from any cause
Overall survival | Assessed from Day 1 throughout the study until individual participant study discontinuation, up to 12 months.
  The time between the first dose date to the date of death from any cause
Number of participants with AEs and SAEs occurring after administration of tocilizumab or etanercept for cytokine release syndrome (CRS) | Throughout study participation, up to 12 months.
Number of participants with changes in cytokines or C-reactive protein after administration of tocilizumab or etanercept | Throughout study participation, up to 12 months.
Outcome of CRS event in participants treated with tocilizumab or etanercept | Throughout study participation, up to 12 months.

CONTACTS AND LOCATIONS:
Overall Officials: Denise Casey, M.D., Study Director — MacroGenics
Locations (7):
- United States (7):
  - Colorado Blood Cancer Network, Denver, Colorado
  - University of Maryland, Greenbaum Comprehensive Cancer Center, Baltimore, Maryland
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - START - Midwest, Grand Rapids, Michigan
  - Washington University School of Medicine, St Louis, Missouri
  - Duke University Medical Center, Durham, North Carolina
  - South Austin Medical Center, Austin, Texas

IPD SHARING:
Plan to Share IPD: No